CLINICAL TRIAL: NCT03537144
Title: Comparison of the Efficacy of IV Acetaminophen Versus IV Indomethacin in Treatment of Hemodynamically Significant PDA in VLBW Infants
Brief Title: Acetaminophen vs Indomethacin in Treating hsPDA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Difficulty enrolling patients
Sponsor: University of Tennessee (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-04411-FB
Record Dates: First submitted 2018-04-30; First posted 2018-05-25 (Actual); Last update posted 2019-12-03 (Actual); Status verified 2018-05

CONDITIONS: Patent Ductus Arteriosus
Keywords: Patent ductus arteriosus; acetaminophen; indomethacin
MeSH Terms: conditions — Ductus Arteriosus, Patent | interventions — Indomethacin; Acetaminophen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Indomethacin (Active Comparator): Indomethacin as drug to treat PDA.
  Interventions: Drug: Indomethacin
- Acetaminophen (Experimental): Acetaminophen as drug to treat PDA.
  Interventions: Drug: Acetaminophen

INTERVENTIONS:
Drug: Indomethacin — IV indomethacin will be given every 12 hours for 3 doses. If <48 hours old, 1st dose 0.2 mg/kg, 2nd dose 0.1 mg/kg, and 3rd dose 0.1mg/kg. If 2-7 days old, 1st dose 0.2 mg/kg, 2nd dose 0.2 mg/kg, and 3rd dose 0.2 mg/kg. If >7 days old, 1st dose 0.2 mg/kg, 2nd dose 0.25 mg/kg, and 3rd dose 0.25 mg/kg.
  Other Names: Indocin
  Arms: Indomethacin
Drug: Acetaminophen — 15mg/kg/dose every 6 hours for 12 doses
  Other Names: Ofirmev
  Arms: Acetaminophen

SUMMARY:
The purpose of this study is to see if acetaminophen (Tylenol) is as effective as indomethacin in closing patent ductus arteriosus in premature infants.

DETAILED DESCRIPTION:
The study will be a randomized, controlled, non-inferiority trial, and the investigators plan to enroll premature infants <32 weeks, <1500g, and who are < 21 days of age at Regional One Health, LeBonheur Children's Hospital, and Methodist Germantown NICUs in Memphis, TN. A study group of 42 patients for each group will be needed to allow a maximum difference of 25% to consider non-inferiority in the closure rate between IV acetaminophen and IV indomethacin (with power of 80% and alpha of 0.05).2 The investigators' goal will be to enroll 50 infants for each treatment group, to help with an expected 20% drop out rate either due to complications or parents removal of consent. Dosages: IV acetaminophen 15mg/kg/dose every 6 hours for 12 doses,6 IV indomethacin dose will depend on age.IV indomethacin will be given every 12 hours for 3 doses. The infants will be eligible for the study after primary attending has made the decision to treat the hsPDA. The goal will be 50 infants in the IV acetaminophen group and 50 infants in the IV indomethacin group.

Informed consent will be obtained from the parent after ECHO has been obtained and the primary attending has decided to treat PDA in the infant who meets inclusion criteria without any of the exclusion criteria. The investigators will use block randomization and stratify by site to generate 140 random values of either 0 for acetaminophen or 1 for indomethacin. The goal will be 50 infants randomized to acetaminophen group and 50 infants randomized to indomethacin group. The numbers will be placed in opaque envelope and opened after consent is obtained. The primary team will not be blinded given the different frequencies of administration of acetaminophen and indomethacin. The first ECHO will be read by staff pediatric cardiologist. A pediatric cardiologist will retrospectively go back and read all ECHOs blinded for standardization.

Prior to induction of treatment, we will record complete blood count (CBC) and complete metabolic panel (CMP) with AST/ALT. After treatment, the investigators will record AST/ALT within 48 hours, and will record follow-up ECHO reports that occur within seven days of initiation of treatment. The decision to repeat treatment will be left to primary attending's discretion. The primary attending will determine any additional medical or surgical treatment if indicated. Data regarding ROP, IVH, and BPD will be collected from patient's chart prior to discharge.

Primary outcome will be the rate of successful PDA treatment by ECHO in each group. Successful PDA treatment will be defined as no longer meeting ECHO criteria for hsPDA. Secondary outcome data will be recorded and include the following: retreatment, surgical closure, days on invasive mechanical ventilation, duration of supplemental oxygen requirement, respiratory support at 36 weeks post-menstrual age (PMA), NEC, ROP, days to full feeds, gastrointestinal perforation, length of stay, renal dysfunction defined by UOP < 1cc/kg/hr in an 8 hour period, creatinine elevation greater than 1.5 mg/dL, and discharge disposition.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age at birth 22 weeks to 31 6/7 weeks.
* Birth weight ≤ 1500 grams
* Day of life ≤ 21 days
* ECHO findings:

Left-to-right ductal flow AND 2 of the following 3:

* Ductal size > 1.5mm at smallest diameter
* Reversal of flow in descending aorta
* Left atrial size to aortic root ratio >1.5
* Platelet count > 50,000

Exclusion Criteria:

* Ductal dependent congenital heart disease
* Major congenital anomaly
* Life-threatening infection
* Urine output < 1cc/kg/hr in prior 8 hours
* Serum creatinine > 1.8 mg/dL
* Hyperbilirubinemia requiring exchange transfusion
* Active NEC Stage 2 or 3 using Bell's staging criteria
* Active intestinal perforation
* Liver dysfunction [2x upper limit of normal for aspartate aminotransferase(AST) and/or alanine aminotransferase (ALT)]
* Active GI bleeding
* Concurrent hydrocortisone use
* Known IVH Grade 3 or 4

Ages: 22 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 37 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Successful treatment of PDA closure | Follow-up ECHO to assess for closure within 7 days of treatment initiation
  Definition of successful treatment of PDA is the PDA no longer meets the echocardiogram inclusion criteria.

SECONDARY OUTCOMES:
PDA retreatment | 1 year
  Did the patient require a second course of treatment with either indomethacin or acetaminophen. Did the PDA require surgical closure.
Supplement O2 requirement at 36 weeks PMA | Until 36 weeks PMA
  Was infant on >21% O2 at 36 weeks post-menstrual age
Nectrotizing enterocolitis | 1 year
  As defined by Bell's Staging criteria, at any time during hospital stay
Gastrointestinal perforation | 1 year
  As defined by xray demonstration of free peritoneal air or as diagnosed by surgery
Mortality | 1 year
  Death before discharge from NICU stay
Days on invasive mechanical ventilation | 1 year
  Days on invasive mechanical ventilation
Days on supplement oxygen | 1 year
  Days on supplement oxygen
Days to full feeds | 1 year
  Day till the infant reaches 120 kcal/kg/d
Length of stay | 1 year
  Time from NICU admission to NICU discharge
Retinopathy of prematurity | 1 year
  Stage of ROP and if any treatment was needed
Creatinine elevation greater than 1.5 mg/dL | 1 year
  Creatinine elevation greater than 1.5 mg/dL

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - LeBonheur Children's Hospital, Memphis, Tennessee
  - Methodist-Lebonheur Germantown Hospital, Memphis, Tennessee
  - Regional One Health, Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Hammerman C, Bin-Nun A, Markovitch E, Schimmel MS, Kaplan M, Fink D. Ductal closure with paracetamol: a surprising new approach to patent ductus arteriosus treatment. Pediatrics. 2011 Dec;128(6):e1618-21. doi: 10.1542/peds.2011-0359. Epub 2011 Nov 7. PMID 22065264
- [Result] Dang D, Wang D, Zhang C, Zhou W, Zhou Q, Wu H. Comparison of oral paracetamol versus ibuprofen in premature infants with patent ductus arteriosus: a randomized controlled trial. PLoS One. 2013 Nov 4;8(11):e77888. doi: 10.1371/journal.pone.0077888. eCollection 2013. PMID 24223740
- [Result] Nadir E, Kassem E, Foldi S, Hochberg A, Feldman M. Paracetamol treatment of patent ductus arteriosus in preterm infants. J Perinatol. 2014 Oct;34(10):748-9. doi: 10.1038/jp.2014.96. Epub 2014 May 22. PMID 24854626
- [Result] Jain A, Shah PS. Diagnosis, Evaluation, and Management of Patent Ductus Arteriosus in Preterm Neonates. JAMA Pediatr. 2015 Sep;169(9):863-72. doi: 10.1001/jamapediatrics.2015.0987. PMID 26168357
- [Result] Oncel MY, Yurttutan S, Degirmencioglu H, Uras N, Altug N, Erdeve O, Dilmen U. Intravenous paracetamol treatment in the management of patent ductus arteriosus in extremely low birth weight infants. Neonatology. 2013;103(3):166-9. doi: 10.1159/000345337. Epub 2012 Dec 19. PMID 23258386
- [Result] EL-Khuffash A, James AT, Cleary A, Semberova J, Franklin O, Miletin J. Late medical therapy of patent ductus arteriosus using intravenous paracetamol. Arch Dis Child Fetal Neonatal Ed. 2015 May;100(3):F253-6. doi: 10.1136/archdischild-2014-307930. Epub 2015 Feb 4. PMID 25653299
- [Result] Gokmen T, Erdeve O, Altug N, Oguz SS, Uras N, Dilmen U. Efficacy and safety of oral versus intravenous ibuprofen in very low birth weight preterm infants with patent ductus arteriosus. J Pediatr. 2011 Apr;158(4):549-554.e1. doi: 10.1016/j.jpeds.2010.10.008. Epub 2010 Nov 20. PMID 21094951
- [Result] Evans N, Malcolm G, Osborn D, Kluckow M. Diagnosis of patent ductus arteriosus in preterm infants. Neonatal Rev 2004; 5: e86-e97.
- [Result] Silverman NH, Lewis AB, Heymann MA, Rudolph AM. Echocardiographic assessment of ductus arteriosus shunt in premature infants. Circulation. 1974 Oct;50(4):821-5. doi: 10.1161/01.cir.50.4.821. No abstract available. PMID 4418268
- [Result] Ellison RC, Peckham GJ, Lang P, Talner NS, Lerer TJ, Lin L, Dooley KJ, Nadas AS. Evaluation of the preterm infant for patent ductus arteriosus. Pediatrics. 1983 Mar;71(3):364-72. PMID 6338474
- [Result] Dash SK, Kabra NS, Avasthi BS, Sharma SR, Padhi P, Ahmed J. Enteral paracetamol or Intravenous Indomethacin for Closure of Patent Ductus Arteriosus in Preterm Neonates: A Randomized Controlled Trial. Indian Pediatr. 2015 Jul;52(7):573-8. doi: 10.1007/s13312-015-0677-z. PMID 26244949
- [Result] Thomson Reuters. Neofax 2011. Montvale, NJ: Thomson Reuters; 2011.
- [Result] Martin, R. J., Fanaroff, A. A., & Walsh, M. C. (2015). Fanaroff and Martin's neonatal-perinatal medicine: Diseases of the fetus and infant (10th ed.). St. Louis, Mo.: Mosby/Elsevier
- [Result] Clyman, R. Patent Ductus Arteriosus in the Preterm Infant. in: C.A. Gleason, SU Devaskar (Eds.) Avery's disease of the newborn.9th ed.WB Saunders, Philadelphia;2012:751-761.
- [Result] Terrin G, Conte F, Oncel MY, Scipione A, McNamara PJ, Simons S, Sinha R, Erdeve O, Tekgunduz KS, Dogan M, Kessel I, Hammerman C, Nadir E, Yurttutan S, Jasani B, Alan S, Manguso F, De Curtis M. Paracetamol for the treatment of patent ductus arteriosus in preterm neonates: a systematic review and meta-analysis. Arch Dis Child Fetal Neonatal Ed. 2016 Mar;101(2):F127-36. doi: 10.1136/archdischild-2014-307312. Epub 2015 Aug 17. PMID 26283668
- [Result] Palmer GM, Atkins M, Anderson BJ, Smith KR, Culnane TJ, McNally CM, Perkins EJ, Chalkiadis GA, Hunt RW. I.V. acetaminophen pharmacokinetics in neonates after multiple doses. Br J Anaesth. 2008 Oct;101(4):523-30. doi: 10.1093/bja/aen208. Epub 2008 Jul 15. PMID 18628265
- [Result] Benitz WE; Committee on Fetus and Newborn, American Academy of Pediatrics. Patent Ductus Arteriosus in Preterm Infants. Pediatrics. 2016 Jan;137(1). doi: 10.1542/peds.2015-3730. Epub 2015 Dec 15. PMID 26672023
- [Result] Gersony WM, Peckham GJ, Ellison RC, Miettinen OS, Nadas AS. Effects of indomethacin in premature infants with patent ductus arteriosus: results of a national collaborative study. J Pediatr. 1983 Jun;102(6):895-906. doi: 10.1016/s0022-3476(83)80022-5. PMID 6343572